CLINICAL TRIAL: NCT02372071
Title: Transcutaneous Bilirubinometry in Neonates With the BiliCare System Compared to the Invasive TSB Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerium Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10003
Record Dates: First submitted 2015-02-22; First posted 2015-02-26 (Estimated); Results first posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: We Will Focus on Assessing the Clinical Performance of the BiliCare Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BiliCare (Other): Two measurements with the BiliCare device
  Interventions: Device: BiliCare

INTERVENTIONS:
Device: BiliCare — Two measurements with the BiliCare device

SUMMARY:
The primary objective of this study is to define the performance evaluation of BiliCare TcB device to the "gold standard" bilirubin tests.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinemia or newborn jaundice impacts over 85% of all newborns [1]. Regardless of the mechanism, excessive hyperbilirubinemia has been traditionally treated with phototherapy to minimize any probable risk of developing bilirubin-induced neurotoxicity. However, earlier and more recent data suggest that pre-discharge bilirubin screening for risk of significant hyperbilirubinemia, whether due to a rapid bilirubin production or an earlier age of onset, has impacted the guidelines for clinical use of phototherapy [1, 2]. In this study, we plan to test the performance of a novel transcutaneous device (BiliCareTM) first for screening for bilirubin levels at postnatal age of 6 to 48 hrs; and possibly also, to substitute the use of this measurement for total plasma/serum bilirubin (TB). This device applies a novel light transmission technology that has the potential to measure bilirubin as a point-of-care test in the subcutaneous tissue, and then uses an internal algorithm to calculate bilirubin levels in the skin. In this proposalstudy, we will to assess the clinical performance of the BiliCare by correlating measurements made by this device to near-concurrent measure of total plasma/serum bilirubin at normative ranges (mean, median, range and inter-quartile ranges ) for all term and late-preterm newborns (including those who are at-risk for jaundice and / or being administered with phototherapy) born to families of diverse race and ethnic backgrounds.

ELIGIBILITY:
Inclusion Criteria:

1. Signed parental informed consent
2. Gestational Age >=24 weeks

Exclusion Criteria:

1. Less than 24 weeks of pregnancy at delivery
2. Bruising at the point of measurement on both ears
3. Birthmarks at the point of measurement on both ears
4. Hematomas at the point of measurement on both ears
5. Excessive Hairiness at the point of measurement on both ears
6. Neonate is during Phototherapy or has been exposed to phototherapy treatment during the last six hours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bar-Oz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Preterm, Late Preterm and Term Newborns: The study population will consist of preterm, late preterm and term newborns (infants >=24 weeks gestational age)
Period: Overall Study
Arm/Group | Preterm, Late Preterm and Term Newborns
Started | 111
Completed | 93
Not Completed | 18
Not completed — Protocol Violation | 18

BASELINE CHARACTERISTICS:
Arm/Group | Preterm, Late Preterm and Term Newborns
Number analyzed (Participants) | 93
Age, Customized [Mean (Standard Deviation); unit: Weeks] — Age ( = Gestational age + Chronological age)
  Weeks
    24<=Gestational Age [weeks]<35 | 33.2 (2.0)
    35<=Gestational Age [weeks] | 38.9 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 48
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White or Tan skin tone)) | 93
  African or Bedouin (Dark Skin tone) | 0

OUTCOME MEASURES:

1. Primary Outcome: BiliCare TcB Result Compared to TSB Result
Time Frame: 30 minutes within taking the blood draw for TSB (either before or after the blood draw)
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- BiliCare TcB Average: The study population will consist of preterm, late preterm and term newborns (infants >=24 weeks gestational age) measured with one BiliCare TcB device without an infection control tip and with one BiliCare TcB device with an infection control tip.
  This is the average of both devices
- Total Serum Bilirubin (TSB): The study population will consist of preterm, late preterm and term newborns (infants >=24 weeks gestational age) measured routinely for total serum bilirubin
Arm/Group | BiliCare TcB Average | Total Serum Bilirubin (TSB)
Number analyzed (Participants) | 93 | 93
mg/dL | 8.0 (4.4) | 7.3 (3.9)

ADVERSE EVENTS:
Arm/Group | Preterm, Late Preterm and Term Newborns
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No